CLINICAL TRIAL: NCT06095232
Title: Pilot Study to Investigate Dietary Changes During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Prof. Dr. Soyoung Q Park, Head of the department Decision making and Nutrition (DNN), German Institute of Human Nutrition
Other Study IDs: Pregnancy and dietary changes
Record Dates: First submitted 2023-08-01; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Menstrual cycle; Nutrition; Cognition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool sample (in order to analyse microbiome data)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Primiparous women will participate in the study during the 1st - 3rd trimester of pregnancy and during the postpartum period.
- Control group: Nulliparous women with a regular natural menstrual cycle will undergo the same study procedure as pregnant women.

SUMMARY:
The aim of this pilot study is to investigate dietary choices and composition during pregnancy and fluctuating sex hormones during the natural menstrual cycle in women. In particular, the investigators are interested in the relationship between diet choice, cognitive performance and diversity of the gut microbiome.

The study will be conducted in a longitudinal/cross-sectional design. Primiparous pregnant women will be investigated during four different time periods (during the 1st-3rd trimester and during the postpartum period). Women with a natural regular menstrual cycle will be assessed during two different hormonal phases of the cycle (early follicular, luteal) and undergo the same study design as pregnant women. Participants will conduct online tasks related to cognitive performance, food approach/avoidance behavior and risk assessment, fill out online questionnaires related to diet, mood, sleep and mental-wellbeing. In addition, participants will log their daily food intake for three days in a food diary and send in a stool sample in order to analyse gut microbiome composition.

DETAILED DESCRIPTION:
Before the beginning of the study, participants will undergo a screening process related to inclusion and exclusion criteria. Upon successful study inclusion the procedure for each study session and both study groups will follow the same order. On Day1 of each time point participants will fill out a browser-based segment which includes questionnaires related to e.g. affect, food intake sleep and cognition (approximately 60 minutes) and are asked to complete four browser-based online tasks including and Approach Avoidance Task, Risk Decision Task, Stop Signal Task, Digit-Substitution Task) (approximately 44 minutes). The app-based segment will be completed during three days (Days 2-4). The timing of this will vary by participant, but takes on average 30 minutes per day for three days. These sessions will take place once each trimester, and once during postpartum. Therefore, each collection period will take approximately 234 minutes (3.9 hours) for a total of ca. 15.6 hours per participant.

The investigators will test the following hypotheses:

H1: Differences in food intake across the course of pregnancy with a decrease in healthy food choices (vegetables, fruits) and an increase in carbohydrates and fat ('high craving' foods) H1.1: Higher intake of fat, carbohydrates during late pregnancy compared to naturally cycling women H1.2: Lower intake of vegetables during late pregnancy compared to naturally cycling women H1.3. Higher Dietary Inflammatory Index (DII) during pregnancy compared to naturally cycling women H2: Better inhibition performance during pregnancy compared to naturally cycling women H2.1: Higher executive functioning/memory predicts healthier food choices (more vegetables/fruits, less fat and sugar intake) H3: Worse food-related memory performance during pregnancy and the postpartum period compared to naturally cycling women H4: Higher implicit food approach tendencies towards 'high craving foods' during pregnancy than the postpartum period and naturally cycling women H4.1: Higher implicit food approach behavior towards 'high craving foods' during late vs. early pregnancy H4.2: Higher implicit food approach behavior is related to food intake of 'high craving foods', carbohydrates, fat H5: Higher risk aversion (less risky choices) during pregnancy compared to naturally cycling women H5.1: Reduction in risky choices higher in early vs. late pregnancy

ELIGIBILITY:
Inclusion Criteria:

* 18-35 year old healthy women
* Primiparous pregnant women experiencing a singleton pregnancy or nulliparous women who have no pregnancy intention within the next year with a regular menstrual cycle (25-35 days) and no use of hormonal contraceptives in the previous 6 months
* Legally competent/Consent to participate
* Language proficiency in German (native speaker, fluent)
* Physically and mentally healthy
* Body mass index (BMI) of 18.5 - 30 kg/m2 (pre-pregnancy)

Exclusion Criteria:

Former or current illnesses of:

* Brain or mind (including anxiety disorders, depression, eating disorders, personality disorders, alcohol, drugs or drug dependence, neurological disorders other than occasional headache, psychiatric or neurological abnormalities)
* Heart or blood circulation/cardiovascular disease (myocardial infarction, stroke, hypertension, hypotension)
* Gastro-intestinal disorders (e.g. colon diseases, irritable bowel syndrome, Crohn's disease)
* endocrine disorders (e.g. thyroid disorders)
* Other serious past or present medical conditions (for example, metabolic syndrome, diabetes).

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Group1: primiparous pregnant women Group2: nulliparous women with a natural menstrual cycle
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2023-08-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Food diary | 3 days during 4 study appointments (in ca. 12 months)
  Changes in dietary composition during pregnancy and the menstrual cycle will be assessed using a food diary. This will allow to analyse food composition based on macronutrients and compare protein, fat and carbohydrate consumption across different time points.
Avoidance/approach behavior (food stimuli, baby vs. adult pictures) | 4 study appointments (in ca. 12 months)
  Participants will undergo an online avoidance approach task in which images are either visually increased or decreased, based on the instruction. In a first trial food images are presented based on craving ratings. The second part consists of pictures of babies and adults assessing possible changes in approach avoidance tendencies to baby stimuli in pregnant women.
Inhibitory control | 4 study appointments (in ca. 12 months)
  Inhibitory control will be assessed using a go/no-go task. Go trials will be presented 80% of the time, in an arrow either pointing towards the right or left is presented. Participants have to respond by pressing either right or left, matching the stimulus presentation. 20% of the time a stop signal (xx) will be presented, requiring no button press from participants.
Risk and decision-making | 4 study appointments (in ca. 12 months)
  Participants will make choices in a lottery task based on risky vs safe options. Risky options are less likely but associated with higher fictional monetary rewards whereas safe options occur with a high likelihood and are associated with less monetary rewards.
Processing speed | 4 study appointments (in ca. 12 months)
  In a digit substitution task, a table with symbols and matching numbers is displayed. For one chosen symbol participants have to indicate the matching symbol as quickly as possible. In order to avoid memory effects, the ordering of symbols and numbers is changed in each trial.

CONTACTS AND LOCATIONS:
Overall Officials: Soyoung Q Park, Prof. Dr., Principal Investigator — German Institute of Human Nutrition
Locations (1):
- German Institute of Human Nutrition, Nuthetal, Brandenburg, Germany